**Statistical Analysis Plan** 

Official Study Title: Guided group telehealth to deliver evidence-based therapeutic care to Black college

students

**NCT Number:** 

**Date of Document:** 03/10/2025

## **Statistical Analysis Plan**

To test the primary hypothesis that participants in the Guided Group Telehealth (GGT) condition will experience reductions in depression and anxiety comparable to those in the Individual Telehealth (IT) condition, we will use a mixed-design repeated measures ANOVA. The within-subjects factor will be time (baseline, week 4, week 8, and week 12), and the between-subjects factor will be therapy condition (GGT vs. IT). The dependent variables will be PHQ-9 and GAD-7 scores, measuring depression and anxiety, respectively. Interaction effects will be examined to assess whether changes in symptom severity over time differ between the two conditions. For secondary analyses, we will use independent samples t-tests to compare user engagement and user experience scores between the two conditions at week 12. Descriptive statistics will be used to summarize engagement data, including participation rates, message frequency, and task completion. Additionally, qualitative analysis will be conducted on open-ended responses from the user experience survey to identify common themes related to participants' satisfaction and perceived effectiveness of the intervention. All analyses will be conducted using an alpha level of 0.05, and effect sizes will be reported alongside p-values. If violations of normality or sphericity are detected, appropriate corrections, such as Greenhouse-Geisser adjustments or nonparametric alternatives, will be applied.